CLINICAL TRIAL: NCT01390974
Title: Bedside Genetic Approach to Identify Clopidogrel CYP2C19 Metabolizer and Optimize Maintenance Thienopyridine Treatment After an Acute Coronary Syndrome: The GAMMA Study
Brief Title: Identification of Clopidogrel CYP2C19 Metabolizer and Thienopyridine Treatment After an Acute Coronary Syndrome
Acronym: GAMMA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: P101203; 2011-A00543-38 (Other: IDRCB)
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS; PCI; thienopyridines; prasugrel therapy; clopidogrel therapy
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated for ACS: ACS patients who recently underwent stent PCI, who are stable and eligible for prasugrel or clopidogrel therapy.

SUMMARY:
To demonstrate that a strategy of fast genetic testing performed in outpatient clinic allows to select adequately one of the 2 antiplatelet treatments approved in the same indication (ACS with PCI - prasugrel 10mg MD or clopidogrel 75mg MD). Patients will reach similar levels of platelet inhibition with the 2 different thienopyridines suggesting optimal risk/benefit ratio in most patients with individualized therapy.

DETAILED DESCRIPTION:
Rationale: There are thresholds of on-treatment platelet reactivity that appear to expose patients either to a risk of thrombotic events (high on-treatment platelet reactivity) or to a risk of bleeding events (low on-treatment platelet reactivity). Clopidogrel is an oral platelet P2Y12 receptor inhibitor that requires metabolic activation catalyzed by several Cytochromes P450 (CYP) isoforms. The loss-of-function polymorphism 2C19*2, carried by 30% of individuals, is associated with high-on-treatment platelet reactivity (low level of P2Y12 inhibition) and a higher risk of stent thrombosis in patients exposed to clopidogrel (OR=3.45 (2.14-5.57)). The gain-of-function polymorphism 2C19*17 is associated with low-on-treatment platelet reactivity (high level of P2Y12 inhibition) with a higher risk of TIMI major bleeding (OR=1.85 (1.19 -2.86). Prasugrel is a new thienopyridine drug with improved ischemic outcomes compared with clopidogrel in acute coronary syndrome patients undergoing PCI but the drug was also associated with more bleeding complications. Prasugrel is a more potent irreversible P2Y12inhibitor than clopidogrel, but it also requires a metabolic conversion that is less or not affected by CYP2C19 variants, unlike clopidogrel. The recent pharmacogenetic literature suggests that individualized treatment (choice between clopidogrel or prasugrel which both are possible in this indication) based on the genetic information rapidly obtained, is possible. This would improve the risk/benefit of therapy. Both common gain- and loss-of function CYP2C19 alleles can be combined to identify two metabolizers status: rapid metabolizer (ultra fast or UF: *17/*17, 5% of all comers and normal metabolizers or NM : *1/*1 et *1/*17, 50% of all comers) at potential higher risk of bleeding and slow metabolizer (Intermediate Metabolizers or IM, *1/*2 and *2/*17, 40% of all comers and Poor Metabolizers or PM, *2/*2, 5% of all comers) at potential higher risk of thrombosis. Primary hypothesis ("genetic hypothesis") : the proportion of rapid metabolizers treated with a 75mg clopidogrel MD within the optimal range of P2Y12 inhibition at 30 days, (defined as a threshold of 220 AU·min up to 350 AU·min of ADP-induced platelet aggregation measured by the Multiple Electrode platelet Aggregometry - Multiplate analyzer, DYNABYTE, Munich, Germany or a % inhibition between 30% up to 80% using the VerifyNowTMP2Y12 platform), is non inferior to the proportion of slow metabolizers treated with prasugrel 10mg MD.Secondary hypothesis ("functional hypothesis"): At 30 days, patients outside the pre-specified target of P2Y12 inhibition level will be adjusted (prasugrel 10mg or clopidogrel 75mg). The hypothesis is that PFT on top of genetic testing will improve the number of patients reaching the prespecified optimal target of P2Y12 inhibition. Thus, the proportion of slow metabolizers within the target at D45 is non inferior to that of rapid metabolizer as determined by the POC PFT. Objectives: To demonstrate that a strategy of fast genetic testing performed in outpatient clinic allows to select adequately one of the 2 antiplatelet treatments approved in the same indication (ACS with PCI - prasugrel 10mg MD or clopidogrel 75mg MD). Patients will reach similar levels of platelet inhibition with the 2 different thienopyridines suggesting optimal risk/benefit ratio in most patients with individualized therapy. Study population: ACS patients who recently underwent stent PCI, who are stable and eligible for prasugrel or clopidogrel therapy.Study design: Prospective,multicenter study. Genetic metabolizer status will be determined using the VerigeneTM (Nanosphere technology) platform during outpatient follow-up visit. Thienopyridine treatment at enrolment will not affect eligibility. Rapid metabolizers (UF and NM) will be treated by 75mg clopidogrel MD while slow metabolizers (IM and PM) will be allocated to prasugrel 10mg MD. A first evaluation of platelet reactivity will be performed one month after to allow the comparison of the proportion of patients who are within the optimal prespecified window of P2Y12 inhibition (primary hypothesis). The investigators will evaluate the hypothesis that a treatment adjustment based on the results obtained by this pharmacodynamic evaluation will improve the rate of success. In this second phase, patients with a level of P2Y12 inhibition >80% (<220AU.min) or <30% (>350 AU.min) will be switched to 75mg clopidogrel MD and or to prasugrel 10mg MD, respectively. A second evaluation of the level of platelet reactivity will be performed at day 45 to allow the comparison of proportions of patients within the prespecified optimal window of P2Y12 inhibition between rapid and slow metabolizer genotypes. Duration of inclusion: 12 months Duration of participation of the patient: 60 days Primary endpoint: Proportion of patient who are within the optimal prespecified window of P2Y12 inhibition at 30 days defined as a threshold of 220 AU·min up to 350 AU·min of ADP-induced platelet aggregation measured by the Multiple Electrode platelet Aggregometry - Multiplate analyzer, DYNABYTE, Munich, Germany or a % inhibition between 30% up to 80% using the VerifyNowTMP2Y12 platform.Number of patients: The investigators have estimated the proportion of prasugrel-treated patients within the prespecified target of P2Y12 inhibition to be 75%. The investigators have formulated the hypothesis that 80% of rapid metabolizers on clopidogrel 75mg MD will stand in the optimal prespecified window of P2Y12 inhibition and the investigators wish to demonstrate that this proportion is not inferior to that of prasugrel-treated patients. Considering a power of 80%, an alpha-risk error of 0.05 and a non-inferiority margin of -10%, a sample size of 122 patients per group are required. Expected results: The GAMMA study will provide answers to a major challenge that is whether rapid genetic information on 2C19 genotype can help in reaching the optimal target of IPA using 2 different thienopyridine, that have different sensitivity to the CYP2C19 variants. Statistical analysis: The non inferiority will be considered as demonstrated (according to the consent risk) if the non inferiority margin of the 95% confidence interval of the difference in percentages is superior to the non inferiority margin (ICH Statistical Procedures). The non-inferiority margin has been established at -10% according to clinical considerations based on an acceptable maximal lost of efficacy.

ELIGIBILITY:
Inclusion Criteria:

- ACS patients who underwent Percutaneous coronary intervention

Exclusion Criteria:

* Anemia <10g/dL
* Indication for VKA
* Recent bleeding or planned surgery
* Thrombopenia <80 000/µl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ACS patients who recently underwent stent PCI, who are stable and eligible for prasugrel or clopidogrel therapy.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
proportion of patients who are within the optimal prespecified window of P2Y12 inhibition | At one month
  the proportion of rapid metabolizers treated with a 75mg clopidogrel MD within the optimal range of P2Y12 inhibition at 30 days, (defined as a threshold of 220 AU·min up to 350 AU·min of ADP-induced platelet aggregation measured by the Multiple Electrode platelet Aggregometry - Multiplate analyzer, Dynabyte, Munich, Germany or a % inhibition between 30% up to 80% using the VerifyNowTMP2Y12 platform),

SECONDARY OUTCOMES:
proportion of patients who are within the optimal prespecified window of P2Y12 inhibition | at 45 days
  the proportion of rapid metabolizers treated with a 75mg clopidogrel MD within the optimal range of P2Y12 inhibition at 30 days, (defined as a threshold of 220 AU·min up to 350 AU·min of ADP-induced platelet aggregation measured by the Multiple Electrode platelet Aggregometry - Multiplate analyzer, Dynabyte, Munich, Germany or a % inhibition between 30% up to 80% using the VerifyNowTMP2Y12 platform),

CONTACTS AND LOCATIONS:
Overall Officials: Jean Philippe COLLET, PUPH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- ACTION-Institut de Cardiologie-Groupe Hospitalier Pitié-Salpêtrière (APHP) Université Pierre et Marie Curie (UPMC), Paris, France